CLINICAL TRIAL: NCT00088894
Title: A Randomized Phase III Trial Of Gemcitabine Plus Bevacizumab (NSC#704865 IND#7621) Versus Gemcitabine Plus Placebo In Patients With Advanced Pancreatic Cancer
Brief Title: Gemcitabine With or Without Bevacizumab in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02960; CALGB-80303; CDR0000377542; U10CA031946 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Bevacizumab; Pharmacogenomic Testing

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (gemcitabine hydrochloride, bevacizumab) (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on days 1 and 15.
  Interventions: Drug: gemcitabine hydrochloride; Biological: bevacizumab; Other: laboratory biomarker analysis; Other: pharmacogenomic studies; Other: pharmacological study
- Arm II (gemcitabine hydrochloride, placebo) (Active Comparator): Patients receive gemcitabine IV as in arm I and placebo IV over 30-90 minutes on days 1 and 15.
  Interventions: Drug: gemcitabine hydrochloride; Other: placebo; Other: laboratory biomarker analysis; Other: pharmacogenomic studies; Other: pharmacological study

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
  Arms: Arm I (gemcitabine hydrochloride, bevacizumab)
Other: placebo — Given IV
  Other Names: PLCB
  Arms: Arm II (gemcitabine hydrochloride, placebo)
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacogenomic studies — Correlative studies
  Other Names: Pharmacogenomic Study
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This randomized phase III trial is studying gemcitabine and bevacizumab to see how well they work compared to gemcitabine alone in treating patients with locally advanced or metastatic pancreatic cancer. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as bevacizumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Bevacizumab may also stop the growth of tumor cells by stopping blood flow to the tumor. Combining gemcitabine with bevacizumab may kill more tumor cells. It is not yet known whether gemcitabine is more effective with or without bevacizumab in treating pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if combination chemotherapy with gemcitabine and bevacizumab achieves superior survival compared to gemcitabine and placebo in patients with previously untreated advanced pancreatic cancer.

SECONDARY OBJECTIVES:

I. To compare the objective response rates, duration of response, progression free survival, and toxicity of these two regimens in patients with advanced pancreatic cancer.

II. To measure baseline levels of VEGF and correlate with treatment outcome. III. To measure baseline and on treatment levels of additional growth factors that may be co- or counter- regulated with VEGF and correlate with response to treatment.

IV. To measure baseline and on treatment levels of coagulation and endothelial cell activation markers that may predict for thrombotic or bleeding risks related to treatment.

V. To generate protein expression profiles using a MALDI-TOF based platform from serum samples. To analyze and compare protein expression profiles to elucidate ion peaks that differentiate patients who respond to therapy from patients who do not respond. To identify proteins responsible for the differentially expressed ion peaks. To develop quantitative assays for each of these proteins.

VI. To assess any differences in overall survival within the treatment arm (gemcitabine + bevacizumab), between the two VEGF genotypic groups: Group 1 denoted by individuals with CT or TT genotypes and Group 2 consisting of individuals with CC genotypes.

VII. To conduct an exploratory analysis of gene-toxicity, gene-response, and gene-survival relationships for the various polymorphisms described in the genes implicated in gemcitabine pharmacology (CDA, DCK, DCTD, SLC29A1, SLC28A1, SLC29A2). An exploratory quantitative interaction between the genotypes (group 1 or 2) and the treatment arms (gemcitabine + bevacizumab or gemcitabine + placebo) in predicting overall survival will also be evaluated.

VIII. To identify specific SNPs and genetic variation that are associated with differences among patients in the risk of toxicity.

IX. To compare the effects of gemcitabine + bevacizumab versus gemcitabine + placebo on resource utilization, cost, and utilities, and if applicable, to make estimates of marginal cost-utility.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to ECOG performance status (0-1 vs 2), disease extent (metastatic vs locally advanced), and prior radiotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on days 1 and 15.

Arm II: Patients receive gemcitabine IV as in arm I and placebo IV over 30-90 minutes on days 1 and 15.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 590 patients (295 per treatment arm) will be accrued for this study within 26.8 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic documentation of adenocarcinoma of the pancreas; documentation of disease extent by CT scan is required; radiologically measurable disease is not required; patients with documented invasion of adjacent organs (e.g., duodenum, stomach) by CT scan are not eligible
* No prior chemotherapy for metastatic disease
* If the patient received adjuvant therapy, it must have been completed at least 4 weeks prior to enrollment on this study; the patient must have recovered from all treatment related toxicities and must have evidence of disease progression following adjuvant treatment
* Prior radiation therapy, with or without a radiosensitizing dose of fluoropyrimidines, is allowed provided the patient has disease outside of the radiation port; at least 4 weeks must have elapsed from completion of the radiation therapy and all signs of toxicity must have resolved
* No prior treatment with gemcitabine or bevacizumab in the adjuvant or metastatic setting
* No current or recent (within 1 month) use of a thrombolytic agent
* Patients may not have had prior therapy with other VEGF inhibitors
* No recent invasive surgical procedures; this includes:

  * Major surgical procedure (e.g. exploratory laparotomy or laparoscopy), open biopsy, or significant traumatic injury within 28 days prior to registration
  * Fine needle aspirations or venous access device within 7 days prior to registration
  * Anticipation of need for major surgical procedures during the course of the study
* No clinically significant cardiovascular disease; this includes:

  * Uncontrolled hypertension (blood pressure > 150/90 on medication)
  * New York Heart Association grade II or greater congestive heart failure
  * Serious cardiac arrhythmia requiring medication
* No recent (within 6 months) arterial thrombotic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina, or myocardial infarction (MI); patients with clinically significant peripheral artery disease (i.e., claudication on less than one block) are also ineligible
* No evidence of CNS disease, including primary brain tumor, or any brain metastasis
* No serious or non-healing wound, ulcer or bone fracture
* No serious active infection (viral, fungal bacterial); no infection requiring parenteral antibiotics at time of registration
* Patients with known hypersensitivity of Chinese hamster ovary cell products or other recombinant human antibodies are not eligible
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers are not to be registered; patients are not considered to have a "currently active" malignancy if they have completed therapy and considered by their physician to be at less than 30% risk of relapse
* Women must be non-pregnant and non-breast feeding
* ECOG Performance status of 0, 1 or 2
* Granulocytes ≥ 1,500/μl
* Platelet count ≥ 100,000/μl
* Creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 60 mL/min
* Total bilirubin ≤ 1 x upper limit of normal
* SGOT(AST) ≤ 2.5 x upper limit of normal
* PT INR =< 1.5, unless patient is on full dose warfarin
* Urine protein; for ≥ 1+ proteinuria, 24 hour urine collection must demonstrate < 1 gm of protein/24 hours
* Required diagnostic procedures:

  * CT of the abdomen
  * Chest x-ray

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2004-06; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From trial entry until death, assessed up to 7 years
  Based on the stratified logrank test.
Discrepancies in the response rate between the two genotypic groups (CT/TT or CC) (Pharmacogenetics portion) | Up to 7 years
  This analysis will be done in the context of a two-way multiplicative logistic model with genotype and treatment as the two factors.
Grade 3-4 neutropenia in terms of specific single-nucleotide polymorphisms (SNPs) and/or copy number variations that are associated with the prevalence of these events (Clinical endpoint) | Up to 7 years

SECONDARY OUTCOMES:
Objective response (complete or partial [CR/PR]) | Up to 7 years
Duration of response | Time from the first tumor assessment that supports the patient's response to the time of disease progression or death from any cause, assessed up to 7 years
Progression-free survival (PFS) | From study entry until documented progression of disease or death from any cause, assessed up to 7 years
  The two-way multiplicative Cox model will be used.
Toxicity graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Up to 7 years
  The two-way multiplicative Cox model will be used.
Quantitative interaction between the genotypes (group 1 or 2) and the treatment arm (gemcitabine or gemcitabine + bevacizumab) in modeling response (Pharmacogenetics portion) | Up to 7 years
Objective response (PR/CR versus stable disease [SD]/progressive disease [PD]) (Clinical endpoint) | Up to 7 years
Disease-control (PR/CR/SD versus PD) (Clinical endpoint) | Up to 7 years
OS (Clinical endpoint) | Up to 7 years
  This endpoint will be analyzed in the framework of a 3x6 singly ordered contingency table.

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States

REFERENCES:
- [Derived] Quintanilha JCF, Wang J, Sibley AB, Jiang C, Etheridge AS, Shen F, Jiang G, Mulkey F, Patel JN, Hertz DL, Dees EC, McLeod HL, Bertagnolli M, Rugo H, Kindler HL, Kelly WK, Ratain MJ, Kroetz DL, Owzar K, Schneider BP, Lin D, Innocenti F. Bevacizumab-induced hypertension and proteinuria: a genome-wide study of more than 1000 patients. Br J Cancer. 2022 Feb;126(2):265-274. doi: 10.1038/s41416-021-01557-w. Epub 2021 Oct 6. PMID 34616010
- [Derived] Quintanilha JCF, Liu Y, Etheridge AS, Yazdani A, Kindler HL, Kelly WK, Nixon AB, Innocenti F. Plasma levels of angiopoietin-2, VEGF-A, and VCAM-1 as markers of bevacizumab-induced hypertension: CALGB 80303 and 90401 (Alliance). Angiogenesis. 2022 Feb;25(1):47-55. doi: 10.1007/s10456-021-09799-1. Epub 2021 May 24. PMID 34028627